CLINICAL TRIAL: NCT05050799
Title: US Post-Market Surveillance Study of the Surfacer* Inside-Out* Access Catheter System (Surfacer System)
Brief Title: US Post-Market Surveillance Study of the Surfacer System
Status: Recruiting | Type: Observational
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CVO-P4-23-01
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Venous Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Central Venous Access — The Surfacer® Inside-Out® Access Catheter System is intended to obtain central venous access to facilitate catheter insertion into the central venous system for patients with upper body venous occlusions or other conditions that preclude central venous access by conventional methods.

SUMMARY:
Single arm, observational, multi-center, consecutively enrolling, post-market surveillance study. Treating patients in need of central venous access who have upper body venous occlusions or other conditions that preclude central venous access by conventional methods, and who meet the requirements described in the device labeling.

DETAILED DESCRIPTION:
Single arm, observational, multi-center, consecutively enrolling, post-market surveillance study. A minimum of 30 patients will be enrolled in the study, all cases to be performed un-proctored at up to 12 sites in the United States, with no site enrolling more than 6 subjects. All patients enrolled will sign an informed consent form for use of their data. Investigators will invite patients who will be treated with the device in accordance with the approved labeling and who met enrollment criteria to join the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have been referred for placement of central venous access, i.e., placement of catheter, nutritional line, etc.
2. Subjects with upper body venous occlusions or other conditions that preclude central venous access by conventional methods
3. Subjects are willing and able to give written informed consent

Exclusion Criteria:

1. Occlusion of the right femoral vein, right iliac vein or inferior vena cava
2. Acute thrombus within any vessel to be crossed by Surfacer System (SVC, jugular, IVC, brachiocephalic and subclavian)
3. Occlusion within the arterial system
4. Occlusion within the coronary or cerebral vasculature

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of central venous access who have upper body venous occlusions or other conditions that preclude central venous access by conventional methods and who meet requirements in the labeling of the IFU.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Central Venous Access operational | 24 hours
  safe insertion of the device to facilitate central venous access
Incidence of adverse events through 24 hours | 24 hours
  no procedural adverse events or peri procedural adverse events

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Pima Heart and Vascular, Tucson, Arizona
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Baylor Scott & White Heart and Vascular Hospital, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Flow Vascular Institute, Pasadena, Texas
  - St. Mark's Hospital, Millcreek, Utah

IPD SHARING:
Plan to Share IPD: No